CLINICAL TRIAL: NCT01064973
Title: An Open Label Extension Study to Evaluate the Safety, Tolerability and Pharmacokinetics of STX209 in Subjects With Autism Spectrum Disorders
Brief Title: An Open Label Extension Study of STX209 in Subjects With Autism Spectrum Disorders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: all active subjects were rolled into study 209AS209/NCT01706523
Sponsor: Seaside Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22007
Record Dates: First submitted 2010-02-05; First posted 2010-02-09 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Autism Spectrum Disorders
Keywords: autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — arbaclofen placarbil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- STX209 (Experimental): STX209 (arbaclofen)
  Interventions: Drug: arbaclofen

INTERVENTIONS:
Drug: arbaclofen — A flexible dose titration will be utilized during the first four weeks to define the optimal titrated dose (OTD) for each subject. Investigators will use clinical judgment to adjust doses to the oral OTD. The starting dose will be 1 mg BID. The dose may be increased every four to five days to 2 mg BID, 3 mg BID, 5 mg BID and then 10 mg BID
  Other Names: R-baclofen, STX209, arbaclofen

SUMMARY:
Study 22003, "An Open-Label, Flexible-Dose Evaluation of the Safety and Tolerability of STX209 for Treatment of Irritability in Subjects With Autism Spectrum Disorders(ASD)" currently is evaluating the efficacy of STX209 (R-baclofen) for management of typical problem behaviors, such as irritability and aggression, in subjects with ASD. This study (22007) will enter subjects who complete Study 22003 into a long-term, open-label study.The open-label extension protocol will provide necessary data on the long-term safety and tolerability of STX209 among subjects with ASD who receive treatment under conditions more closely reflective of their general medical care.

ELIGIBILITY:
Inclusion Criteria:

* Have completed all scheduled visits in protocol 22003 and have shown they can adequately follow the protocol, with sufficient medical justification to continue on open-label treatment with STX209, as assessed by the principal investigator

Exclusion Criteria:

* Subjects with a medical condition that might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being.
* The occurrence or continuation of any adverse event or condition during study 22003 that, in the opinion of the Investigator, should exclude the subject from participating in this open-label extension

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Irritability subscale of the Aberrant Behavior Checklist | every 2 to 3 months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - University of California-Los Angeles Neuropsychiatric Institute, Los Angeles, California
  - Yale Child Study Center, New Haven, Connecticut
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of North Carolina Neurosciences Hospital, Chapel Hill, North Carolina
  - Vanderbilt Kennedy Center, Nashville, Tennessee
  - Red Oaks Psychiatry Associates, P.A., Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington